CLINICAL TRIAL: NCT02913833
Title: The Impact of Pain Assessment on the Hospital Length of Stay of Patients in a Rehabilitation Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Samar Hatem, Head of clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUB- EVA-REVA
Record Dates: First submitted 2016-09-15; First posted 2016-09-26 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Pain
Keywords: Pain; Hospital length of stay; Revalidation unit
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily pain evaluation (Experimental): Patients recruited in a sequential order within the chronic revalidation unit of the CHU Brugmann hospital, Queen Astrid site.
  Interventions: Other: Pain evaluation
- Control (No Intervention): Patients recruited in a sequential order within the chronic revalidation unit of the CHU Brugmann hospital, Queen Astrid site.

INTERVENTIONS:
Other: Pain evaluation — Pain will be assessed four times per day on a visual analogic scale.
  Arms: Daily pain evaluation

SUMMARY:
The financing of the Belgian hospitals is based on a system taking into account the length of hospitalization of a given patient according to his/her pathology, his/her age and his/her geriatric characteristics. This system encourages all hospital to lower the hospitalization duration to the national average for these criteria. This results in better efficiency in the management of hospitalizations but also means a swifter transfer to structures exempted from this system such as revalidation units, nursing homes and psychiatric units. An assessment of the differences in the medical practice, in terms of quality and outcomes of care, is essential for any reform willing to reduce medical costs.

Pain management is part of the quality indicators within hospitals. Pain is defined by the International Association for the Study of Pain as "an unpleasant sensory and emotional experience, associated to present or potential tissue damage, or described in terms of such a damage". Several studies have showed that pain affects the quality of life and impacts the daily activities. Acute or chronic pain can cause adverse symptoms such as sleep disturbance, appetite loss, decreased concentration, mood changes and the disruption of familial, work and social activities. Pain might also slow down revalidation processes. A study performed by Aprile et al showed that pain negatively influenced the rehabilitation program of a quarter of the patients having had a stroke. The functional recovery was slower and the costs were higher.

The aim of this study is to determine if the systematic evaluation of the pain of a patient hospitalized in a revalidation unit has an impact on his/her length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Sequential inclusion of all patients hospitalized in the chronic revalidation hospital unit of the CHU Brugmann - Queen Astrid site

Exclusion Criteria:

* Pathological cognitive state (MMS<23/30)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Pain score (EVA) | 5 minutes, 4 times per day
  Pain assessment on the Visual Analogic Scale (EVA)
Hospitalization duration | Hospitalization length (average of 48 days)
HADS score | Baseline (first day of hospitalisation)
  Hospital Anxiety Depression Scale (questionnaire)
HADS score | Day 30 of hospitalisation
  Hospital Anxiety Depression Scale (questionnaire)
Barthel Index | Baseline (first day of hospitalisation)
  Daily life activities assessment
Barthel Index | Day 30 of hospitalisation
  Daily life activities assessment
CACS score | Hospitalization length (average of 48 days)
  Composite score of analgesics consumption

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aprile I, Briani C, Pazzaglia C, Cecchi F, Negrini S, Padua L; Don Carlo Gnocchi Pain-Rehab Group. Pain in stroke patients: characteristics and impact on the rehabilitation treatment. A multicenter cross-sectional study. Eur J Phys Rehabil Med. 2015 Dec;51(6):725-36. Epub 2015 Feb 26. PMID 25739508
- [Background] Kreling MC, da Cruz DA, Pimenta CA. [Prevalence of chronic pain in adult workers]. Rev Bras Enferm. 2006 Jul-Aug;59(4):509-13. doi: 10.1590/s0034-71672006000400007. Portuguese. PMID 17340726
- [Background] Schoenthaler M, Miernik A, Offner K, Karcz WK, Hauschke D, Sevcenco S, Kuehhas FE, Bach C, Buchholz N, Wilhelm K. The cumulative analgesic consumption score (CACS): evaluation of a new score to describe postsurgical analgesic consumption as a surrogate parameter for postoperative pain and invasiveness of surgical procedures. Int Braz J Urol. 2014 May-Jun;40(3):330-6. doi: 10.1590/S1677-5538.IBJU.2014.03.06. PMID 25010299